| Official Title of the Study: |
|---|
| Graphene-Reinforced CAD/CAM Restorations for MIH-Affected Molars in Adolescents: A |
| Prospective Clinical Study |
| NCT Number: |
| NCT: Not yet assigned |
| Document Type: |
| Study Protocol |
| Document Date: |
| December 11th, 2025 |
| Version: |
| 3.0 |
| Sponsor: |
| Universitat Internacional de Catalunya (UIC) |
| Study Sites: |
| Universitat Internacional de Catalunya — Department of Restorative Dentistry |
| University of Barcelona |

# 1. BACKGROUND AND SCIENTIFIC RATIONALE

Molar–Incisor Hypomineralization (MIH) is a qualitative enamel defect affecting 10–20% of European children. MIH molars show porosity, post-eruptive breakdown, and hypersensitivity, reducing the predictability of conventional restorative treatments. Current therapy options—composites, resin-modified glass ionomers, stainless-steel crowns—face limitations such as polymerization shrinkage, marginal degradation, and short service life.

Advances in nanotechnology have introduced graphene-based biomaterials featuring high flexural strength (>180 MPa), biocompatibility, and favorable esthetics. Graphene-reinforced CAD/CAM polymers (e.g., G-CAM®) permit minimally invasive adhesive restorations that may improve outcomes in MIH-affected posterior teeth.

This study prospectively evaluates the 12-month clinical performance of graphene-reinforced CAD/CAM indirect restorations in adolescent MIH patients.

# 2. STUDY OBJECTIVES AND HYPOTHESIS

## **Primary Hypothesis**

Graphene-reinforced CAD/CAM indirect restorations provide high clinical acceptability at 12 months, according to predefined FDI criteria, while reducing postoperative hypersensitivity relative to baseline and preserving structural tooth integrity.

## **Primary Objective**

Evaluate the overall clinical performance of graphene-reinforced CAD/CAM inlays/onlays/overlays in MIH-affected molars at 12 months.

### **Secondary Objectives**

- Assess FDI domain scores: marginal integrity, surface roughness, color stability, fractures, proximal contacts, occlusion/function, and soft-tissue response.
- Measure postoperative sensitivity using VAS.
- Assess patient-reported satisfaction.
- Evaluate structural preservation via pre/post 3D scans.
- Measure restoration survival (Kaplan–Meier).
- Assess workflow efficiency (chair time, need for adjustments).

# 3. STUDY DESIGN

A prospective, single-arm, monocentric, interventional clinical study with 12-month follow-up.

**Number of participants:** 30 adolescents (10–16 years old).

Study duration: 18 months.

# 4. STUDY POPULATION

### **Inclusion Criteria**

- Adolescents aged 10–16.
- Permanent molars with moderate/severe MIH (EAPD).
- Vital, restorable teeth.
- Ability to attend follow-ups.• Informed consent + minor assent.

#### **Exclusion Criteria**

- Fluorosis, amelogenesis imperfecta, other enamel anomalies.
- Severe bruxism.
- Extensive active caries or irreversible pulpitis.
- Systemic diseases affecting enamel/healing.
- Allergy to dental materials.
- Analgesics/AINE <24 h before baseline sensitivity assessment.

# 5. STUDY INTERVENTION

All participants undergo:

- 1. Baseline diagnostics and imaging
- 2. Minimally invasive cavity preparation
- 3. Composite base build-up if required
- 4. CAD/CAM fabrication of graphene-reinforced polymer inlay/onlay/overlay
- 5. Adhesive cementation under rubber dam
- 6. Finishing and occlusal evaluation

Material used: Graphene-reinforced CAD/CAM polymer block (G-CAM®)

# 6. OUTCOME MEASURES

### **Primary Outcomes**

- 1. FDI Global Acceptability (Success = all domains ≤3) at 12 months
- 2. Postoperative sensitivity (VAS 0–10) at baseline, 48 h, 1, 3, 6, 12 months

### **Secondary Outcomes**

- Patient satisfaction (Likert 1–5)
- Structural preservation (volumetric analysis of 3D scans)
- Vitality retention

- Restoration survival (Kaplan–Meier)
- Workflow efficiency (chair time, adjustments)

## 7. SAFETY AND ADVERSE EVENTS

Adverse events include:

- Persistent pain >72 h
- Severe hypersensitivity (VAS ≥7)
- Soft-tissue inflammation
- Partial or total restoration failure
- Complications requiring reintervention

# 8. DATA COLLECTION AND MANAGEMENT

- Standardized photos and 3D scans at baseline and follow-up.
- Pseudonymized data stored on encrypted servers at Dental Esthetic BCN, GDPR compliant.
- Data preserved 15 years, then securely destroyed.• Investigator and promoter maintain separate encrypted linkage file.

# 9. STATISTICAL ANALYSIS PLAN (SAP)

## Sample Size

30 participants (27 required for detecting a  $\geq$ 2-point VAS reduction;  $\beta$ =0.80,  $\alpha$ =0.05).

### **Analysis Methods**

### **Descriptive Statistics**

Mean  $\pm$  SD, median [IQR], and proportions.

### **Primary Analyses**

• FDI scores (ordinal):

Friedman repeated-measures test + Holm correction or ordinal mixed-effects model (time = fixed, participant = random)

• VAS sensitivity (continuous):

Linear mixed-effects model or repeated-measures ANOVA (Greenhouse-Geisser correction)

### **Survival Analysis**

- Kaplan–Meier survival curve
- Failure = debonding or fracture requiring replacement

### **Performance Threshold Tests**

- FDI success proportion at 12 months with 95% CI
- One-sample binomial test vs threshold ≥80%
- Mean VAS reduction ≥2 points with CI>0

### **Missing Data**

- Missing-at-random assumption
- Mixed models inherently robust; no imputation planned

### **Interim Analysis**

None planned.

# 10. ETHICAL CONSIDERATIONS

- Conducted under the Declaration of Helsinki and GDPR.
- CEIm HOUB approval granted (protocol version 3.0).
- Informed consent from guardian + patient assent.
- No biological samples collected.
- Minimal risk: all materials CE-marked and used in routine care.

# 11. ADMINISTRATIVE INFORMATION

**Study Site:** 

Dental Esthetic BCN

**Funding:** 

Self-funded (material costs detailed in protocol).